CLINICAL TRIAL: NCT02779855
Title: A Phase 1/2 Study of Talimogene Laherparepvec in Combination With Neoadjuvant Chemotherapy in Triple Negative Breast Cancer
Brief Title: Talimogene Laherparepvec in Combination With Neoadjuvant Chemotherapy in Triple Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18621
Record Dates: First submitted 2016-05-19; First posted 2016-05-20 (Estimated); Results first posted 2021-10-28 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Ductal Carcinoma; Invasive Breast Carcinoma; Invasive Ductal Breast Carcinoma
Keywords: triple negative breast cancer (TNBC); estrogen receptor; progesterone receptor; invasive ductal carcinoma; breast cancer tumors
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal; Carcinoma, Ductal, Breast; Triple Negative Breast Neoplasms | interventions — talimogene laherparepvec; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Talimogene laherparepvec + Chemotherapy (Experimental): Talimogene laherparepvec with Neoadjuvant Paclitaxel Chemotherapy treatment administration on an outpatient basis. Phase I: Dose Escalation to Determine Maximum Tolerated Dose (MTD). Phase II: Treatment at MTD.
  Interventions: Biological: Talimogene laherparepvec; Drug: Paclitaxel

INTERVENTIONS:
Biological: Talimogene laherparepvec — Talimogene laherparepvec injection. Phase I: Dose escalation. Phase II: Treatment at Maximum Tolerated Dose (MTD) from Phase I. The MTD dose level is defined as the highest dose level with ≤1 out of 6 patients experiencing a dose limiting toxicity (DLT).
  Other Names: IMLYGIC™; modified herpes simplex 1 virus
Drug: Paclitaxel — Paclitaxel chemotherapy infusion. The paclitaxel weekly dose is fixed at 80 mg/m^2.
  Other Names: Taxol®

SUMMARY:
The purpose of this study is to determine if an oncolytic virus called Talimogene laherparepvec (a modified herpes simplex 1 virus that can specifically destroy cancer cells while leaving normal cells alone) injected directly into the tumor during chemotherapy prior to surgery can enhance the elimination of triple negative breast cancer tumors. The natural herpes simplex 1 virus typically causes cold sores around the mouth, but the talimogene laherparepvec version of the herpes virus has been changed to prevent it from reproducing in normal tissue.

However, it can still attack and break open cancer tissue which is why it is used as a treatment for cancer. It is thought that this virus can also help recruit the participant's immune system to attack the cancer cells during their treatment and possibly destroy the tumor tissue more effectively than chemotherapy alone. This virus is already FDA approved to treat melanoma skin tumors, so investigators want to determine if this virus can achieve a similar benefit in women with triple negative breast tumors.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed clinical stage T2-3 N0-2 triple negative (estrogen receptor/progesterone receptor <1% human epidermal growth factor receptor 2 (HER2) 0-1 by ImmunoHistoChemistry (IHC) or unamplified by fluorescence in situ hybridization (FISH)) invasive ductal carcinoma.
* Must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. As well, participants must have primary tumor able to be visualized on ultrasound and amenable to direct injection.
* No prior history of an invasive breast cancer
* Adults ages 18-70
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Must have normal organ and marrow function as outlined in protocol
* Sexually active women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* T4 tumors, known metastatic disease, recurrent disease, inflammatory breast cancer, multicentric disease, and/or synchronous bilateral breast cancer
* A second active malignancy, exceptions are localized non-melanoma skin cancers or prior in situ carcinoma
* Receiving any other investigational agents or are unable to be treated with doxorubicin, cyclophosphamide, and paclitaxel.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to talimogene laherparepvec or other agents used in the study
* Known active or prior herpes simplex virus infections (HSV), prior complications from HSV infections such as encephalitis, or require systemic antiviral therapy at the time of study enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, known active hepatitis B/C infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women who are pregnant or nursing
* Immunocompromised patients may be at increased risk of herpetic infections when treated with talimogene laherparepvec. Therefore, HIV-positive patients, patients with acquired or congenital immunodeficiency conditions, those on chronic systemic immunosuppressants (requiring > 10 mg of prednisone or equivalent/day), Those with active autoimmune disease are excluded from the study.
* Have received any live vaccine therapies used for the prevention of infectious disease within 28 days prior to enrollment and during treatment period. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed. However, intranasal influenza vaccines (eg, Flu - Mist®) are live attenuated vaccines, and are not allowed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2026-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Soliman, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Soliman H, Hogue D, Han H, Mooney B, Costa R, Lee MC, Niell B, Williams A, Chau A, Falcon S, Soyano A, Armaghani A, Khakpour N, Weinfurtner RJ, Hoover S, Kiluk J, Laronga C, Rosa M, Khong H, Czerniecki B. Oncolytic T-VEC virotherapy plus neoadjuvant chemotherapy in nonmetastatic triple-negative breast cancer: a phase 2 trial. Nat Med. 2023 Feb;29(2):450-457. doi: 10.1038/s41591-023-02210-0. Epub 2023 Feb 9. PMID 36759673
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Groups:
- Talimogene Laherparepvec + Chemotherapy -Phase 1 Dose Level 1: Talimogene laherparepvec with Neoadjuvant Paclitaxel Chemotherapy treatment administration on an outpatient basis. Phase I Dose Level 1: 10^6 PFU (plaque forming units) for all five injections
  Paclitaxel: Paclitaxel chemotherapy infusion. The paclitaxel weekly dose is fixed at 80 mg/m^2.
- Talimogene Laherparepvec + Chemotherapy -Phase 1 Dose Level 2: Talimogene laherparepvec with Neoadjuvant Paclitaxel Chemotherapy treatment administration on an outpatient basis. Phase I Dose Level 2: 10^6 PFU (plaque forming units) 1st injection, followed by 10^8 for remaining injections
  Paclitaxel: Paclitaxel chemotherapy infusion. The paclitaxel weekly dose is fixed at 80 mg/m^2.
- Talimogene Laherparepvec + Chemotherapy -Phase 2: Talimogene laherparepvec with Neoadjuvant Paclitaxel Chemotherapy treatment administration on an outpatient basis. Phase 2 at MTD
  Paclitaxel: Paclitaxel chemotherapy infusion. The paclitaxel weekly dose is fixed at 80 mg/m^2.
Period: Overall Study
Arm/Group | Talimogene Laherparepvec + Chemotherapy -Phase 1 Dose Level 1 | Talimogene Laherparepvec + Chemotherapy -Phase 1 Dose Level 2 | Talimogene Laherparepvec + Chemotherapy -Phase 2
Started | 4 | 6 | 40
Completed | 3 | 6 | 40
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by patient prior to treatment | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1 Dose Level 1: Talimogene laherparepvec with Neoadjuvant Paclitaxel Chemotherapy treatment administration on an outpatient basis. Phase I Dose Level 1: 10^6 PFU (plaque forming units) for all five injections
  Paclitaxel: Paclitaxel chemotherapy infusion. The paclitaxel weekly dose is fixed at 80 mg/m^2.
- Phase 1 Dose Level 2: Talimogene laherparepvec with Neoadjuvant Paclitaxel Chemotherapy treatment administration on an outpatient basis. Phase I Dose Level 2: 10^6 PFU (plaque forming units) 1st injection, followed by 10^8 for remaining injections.
  Paclitaxel: Paclitaxel chemotherapy infusion. The paclitaxel weekly dose is fixed at 80 mg/m^2.
- Phase 2: Phase II: Treatment at Maximum Tolerated Dose (MTD) from Phase I. The MTD dose level is defined as the highest dose level with ≤1 out of 6 patients experiencing a dose limiting toxicity (DLT).
  Talimogene laherparepvec: Talimogene laherparepvec injection. Phase II: treatment at MTD
  Paclitaxel: Paclitaxel chemotherapy infusion. The paclitaxel weekly dose is fixed at 80 mg/m^2.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 2 | Total
Number analyzed (Participants) | 3 | 6 | 40 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 38 | 47
  >=65 years | 0 | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 40 | 49
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 6 | 10
  Not Hispanic or Latino | 1 | 4 | 33 | 38
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 4 | 6
  White | 2 | 3 | 27 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 40 | 49

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) / Recommended Phase II Dose (RP2D)
Description: MTD/RP2D of talimogene laherparepvec administered with neoadjuvant paclitaxel- doxorubicin/cyclophosphamide chemotherapy.
Time Frame: Up to 6 months
Measure: Number; unit: million plaque forming units per mL
Arm/Group | Talimogene Laherparepvec + Chemotherapy
Number analyzed (Participants) | 9
million plaque forming units per mL | 100

2. Primary Outcome: Phase II: Percentage of Participants With Pathologic Complete Response Rate (pCR)
Description: Perceptage of participants with pCR following study treatment, defined as: Disappearance of histopathologic evidence of malignant cells in breast and axillary lymph nodes.
Time Frame: Up to 36 months
Population: All patients evaluable for response per protocol
Measure: Number; unit: percentage of participants
Groups:
- Phase 1 Dose Level 2: Talimogene laherparepvec with Neoadjuvant Paclitaxel Chemotherapy treatment administration on an outpatient basis. Phase I Dose Level 2: 10^6 PFU (plaque forming units) 1st injection, followed by 10^8 PFU for remaining injections.
  Paclitaxel: Paclitaxel chemotherapy infusion. The paclitaxel weekly dose is fixed at 80 mg/m^2.
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 2
Number analyzed (Participants) | 3 | 6 | 37
percentage of participants | 66.7 | 50 | 43.24

3. Other Pre Specified Outcome: Recurrence Free Survival Rate
Description: Percentage of participants who are disease recurrence free at 5 year follow-up.
Time Frame: Up to 5 years follow-up
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Overall Survival (OS) Rate
Description: Percentage of participants who are alive at 5 year follow-up.
Time Frame: Up to 5 years follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events collected from on study date to 30 days post last study treatment (3 years, 4.5 months)
Groups:
- Phase 1 Dose Level 1: .Talimogene laherparepvec with Neoadjuvant Paclitaxel Chemotherapy treatment administration on an outpatient basis. Phase I Dose Level 1: 10^6 PFU (plaque forming units) for all five injections
  Paclitaxel: Paclitaxel chemotherapy infusion. The paclitaxel weekly dose is fixed at 80 mg/m^2.
- Phase 1 Dose Level 2: .Talimogene laherparepvec with Neoadjuvant Paclitaxel Chemotherapy treatment administration on an outpatient basis. Phase I Dose Level 1: 10^6 PFU (plaque forming units) 1st injection, followed by 10^8 PFU for remaining injections.
  Paclitaxel: Paclitaxel chemotherapy infusion. The paclitaxel weekly dose is fixed at 80 mg/m^2.
- Phase 2: Phase II: Treatment at Maximum Tolerated Dose (MTD) . The MTD dose level is defined as the highest dose level with ≤1 out of 6 patients experiencing a dose limiting toxicity (DLT).
  Talimogene laherparepvec: Talimogene laherparepvec injection. Phase II: treatment at MTD
  Paclitaxel: Paclitaxel chemotherapy infusion. The paclitaxel weekly dose is fixed at 80 mg/m^2.
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 4/6 | 1/40
Serious Adverse Events (participants affected / at risk) | 1/3 | 4/6 | 7/40
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 (N=3) | Phase 1 Dose Level 2 (N=6) | Phase 2 (N=40)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (3) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 3 (3)
Periorbital infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neuropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 (N=3) | Phase 1 Dose Level 2 (N=6) | Phase 2 (N=40)
Fatigue (General disorders) | 1 (2) | 4 (9) | 34 (59)
Fever (General disorders) | 3 (4) | 5 (6) | 18 (37)
Chills (General disorders) | 0 (0) | 3 (4) | 21 (37)
Flu like symptoms (General disorders) | 2 (2) | 3 (3) | 10 (15)
Injection site reaction (General disorders) | 1 (3) | 3 (4) | 10 (15)
Infusion related reaction (General disorders) | 2 (4) | 4 (5) | 7 (13)
Pain (General disorders) | 0 (0) | 2 (2) | 10 (11)
Edema limbs (General disorders) | 1 (1) | 2 (3) | 9 (13)
Non-cardiac chest pain (General disorders) | 0 (0) | 4 (4) | 4 (5)
Edema face (General disorders) | 0 (0) | 0 (0) | 3 (3)
Malaise (General disorders) | 0 (0) | 1 (1) | 2 (2)
General disorders and administration site conditions - Other (General disorders) | 1 (1) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Neck edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (16) | 6 (26) | 35 (102)
Leukocystosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (7)
Febrile neuropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Blood and lymphatic system disorders -Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (4) | 6 (12) | 29 (51)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 16 (29)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 15 (18)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 3 (3) | 14 (17)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 3 (5) | 9 (10)
Vomitting (Gastrointestinal disorders) | 1 (1) | 4 (6) | 9 (13)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 11 (19)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 11 (12)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (3) | 4 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 18 (23)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 14 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5) | 13 (14)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 6 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 5 (5)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 5 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (6)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 4 (4)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 5 (5)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (5) | 5 (11) | 19 (43)
Alanine aminotransferase increased (Investigations) | 1 (2) | 4 (7) | 17 (26)
Neutrophil count decreased (Investigations) | 1 (3) | 5 (10) | 16 (51)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 13 (15)
Platelet count decreased (Investigations) | 1 (1) | 2 (2) | 7 (10)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (4) | 6 (6)
Weight gain (Investigations) | 0 (0) | 1 (2) | 4 (4)
Weight loss (Investigations) | 0 (0) | 0 (0) | 5 (6)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 3 (8) | 25 (38)
Headache (Nervous system disorders) | 2 (3) | 2 (4) | 20 (33)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 11 (15)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 12 (14)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 13 (18)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 10 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (5)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 12 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 10 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 12 (19)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 8 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 5 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 4 (5) | 13 (16)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 10 (15)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 5 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 6 (12)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1) | 4 (4)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (5)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 4 (6)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Papulopustular rash (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Periorbital infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 15 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 9 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 10 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 6 (6)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (5)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Hot flashes (Vascular disorders) | 1 (1) | 2 (2) | 6 (6)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 7 (10)
Hematoma (Vascular disorders) | 1 (1) | 2 (3) | 3 (3)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 4 (5)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 7 (9)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 6 (6)
Eye disorders - Other (Eye disorders) | 0 (0) | 0 (0) | 4 (6)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 4 (5)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Papilledema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 7 (9)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 4 (6)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (4)
Confusion (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 9 (14)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 3 (3)
Vascular access complication (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 4 (4)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 4 (6)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 3 (4)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1) | 5 (5)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (3)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Menopause (Social circumstances) | 2 (2) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT02779855/Prot_SAP_000.pdf